CLINICAL TRIAL: NCT01034293
Title: Effect of Feeding Frequency on Glucose and Insulin Metabolism and Substrate Partitioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Nederlandse Zuivel Organisatie (Other)
Responsible Party: Prof. dr. WHM Saris, University of Maastricht
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MEC 09-3-032
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Insulin; Glucose Metabolism
Keywords: feeding frequency; insulin metabolism; glucose metabolism; substrate partitioning
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- low feeding frequency (3x) (Experimental)
  Interventions: Dietary Supplement: low feeding frequency (3x)
- High feeding frequency (14x) (Experimental)
  Interventions: Dietary Supplement: High feeding frequency (14x)

INTERVENTIONS:
Dietary Supplement: low feeding frequency (3x) — 3 meals a day
  Arms: low feeding frequency (3x)
Dietary Supplement: High feeding frequency (14x) — 14 meals a day
  Arms: High feeding frequency (14x)

SUMMARY:
The purpose of this study is to determine the effect of feeding frequency on glucose and insulin metabolism and substrate partitioning.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18.5-25 kg/m2 (lean)
* Gender: Male
* Age: subjects has to be older than 18 and including 35 years old
* Caucasian

Exclusion Criteria:

* Metabolic abnormalities such as:

  1. Lactose intolerant
  2. Diabetes Mellitus
  3. Hypertension
  4. Hypotension
  5. Cardiovascular diseases
  6. Asthma and other obstructive pulmonary diseases
  7. Elevated fasting blood glucose level

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Glucose and insulin metabolism | 24 h

SECONDARY OUTCOMES:
Substrate partitioning and metabolic markers | 24 h

CONTACTS AND LOCATIONS:
Overall Officials: WHM Saris, Prof. Dr., Principal Investigator — Maastricht University
Locations (1):
- University of Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Munsters MJ, Saris WH. Effects of meal frequency on metabolic profiles and substrate partitioning in lean healthy males. PLoS One. 2012;7(6):e38632. doi: 10.1371/journal.pone.0038632. Epub 2012 Jun 13. PMID 22719910